CLINICAL TRIAL: NCT04419571
Title: Emergency Laparotomies and Outcomes During the COVID-19 Pandemic - a Retrospective Cohort Study
Brief Title: Outcomes in Emergency Laparotomies During COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Barking, Havering and Redbridge University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Nader Habib Bedwani, Doctor, Barking, Havering and Redbridge University Hospitals NHS Trust
Other Study IDs: 133196
Record Dates: First submitted 2020-06-04; First posted 2020-06-05 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: COVID-19; Emergency General Surgery
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Suspected or Confirmed COVID-19: All adult patients (>17 years) undergoing emergency (laparotomy) surgery at a single centre (Queens Hospital, Romford, UK) with clinically or radiologically suspected COVID-19, or with viral PCR confirmation; diagnosis made 7-days before and 30-days after date of surgery in accordance with the COVIDsurg study criteria (3).
  Interventions: Procedure: Emergency Laparotomy
- Negative or non-suspected COVID-19: All adult patients (>17 years) undergoing emergency (laparotomy) surgery at a single centre (Queens Hospital, Romford, UK) without clinically or radiologically suspected COVID-19, or without viral PCR (Polymerase Chain Reaction) confirmation.
  Interventions: Procedure: Emergency Laparotomy

INTERVENTIONS:
Procedure: Emergency Laparotomy — All adult patients undergoing emergency laparotomy

SUMMARY:
NLR has previously been observed to correlate with complications in upper GI (1) and colorectal (2) surgery. The investigators sought to assess if a similar correlation can be identified in emergency general surgical patients and if the presence of suspected or confirmed COVID-19 may impact on this.

Given the heterogeneity of emergency general surgery the investigators therefore plan to perform a retrospective review of patients having emergency laparotomies only at a single NHS site during COVID-19 pandemic. Assessment of outcomes and Neutrophil:lymphocyte ratio as a predictor of outcomes will be completed. Outcomes will be completed in line with the recent COVIDSurg study criteria (3). The primary outcome is 30-day mortality. Secondary outcomes are 7-day mortality, re-operation, length of stay, post-operative respiratory failure, post-operative ARDS (Acute Respiratory Distress Syndrome), post-operative sepsis and ITU (Intensive Therapy Unit)/HDU (High Dependency Unit) admission.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing emergency laparotomy (change made due to heterogeneity of emergency general surgery)

Exclusion Criteria:

* Inherited or acquired immunodeficiency (which may directly skew NLR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult patients (>17 years) undergoing emergency (laparotomy) surgery at a single centre (Queens Hospital, Romford, UK) regardless of COVID-19 status will be included.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  Mortality

SECONDARY OUTCOMES:
7-day mortality | 7 days
  Mortality
Number of participants returning to theatre | 30 days
  Re-operation
Length of stay | 30 days
  Inpatient stay during index admission
Post-operative respiratory failure | 30 days
  Presence of respiratory failure in the post-operative period as defined in the clinical notes or discharge summaries
Post-operative ARDS | 30 days
  ARDS diagnosed radiologically
Post-operative sepsis | 30 days
  Presence of sepsis in the post-operative period as defined in the clinical notes or discharge summaries
ITU/HDU admission | 30 days
  ITU/HDU admission post-operatively

OTHER OUTCOMES:
Other complications | 30 days
  Other documented post-operative complications
Peri-operative NLR | First 3 post-operative days
  Neutrophil:Lymphocyte Ratio will be recorded daily in the peri-operative period
Post-operative platelet counts | First 3 post-operative days
  Absolute platelet counts recorded daily in the peri-operative period
Post-operative coagulopathy | First 3 post-operative days
  Defined as the presence of increased PT (prothrombin time) OR APTT (activated partial thromboplastin time) OR TT (thrombin time) OR fibrinogen above 1.5X the upper limit of normal. Coagulation will either be defined as normal or abnormal for each patient if one or more of these derangement are identified.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's Hospital, Romford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD regardless of inclusion in final publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available from completion of study for 10 years
Access Criteria: On request

REFERENCES:
- [Background] Vulliamy P, McCluney S, Mukherjee S, Ashby L, Amalesh T. Postoperative Elevation of the Neutrophil: Lymphocyte Ratio Predicts Complications Following Esophageal Resection. World J Surg. 2016 Jun;40(6):1397-403. doi: 10.1007/s00268-016-3427-z. PMID 26813540
- [Background] Cook EJ, Walsh SR, Farooq N, Alberts JC, Justin TA, Keeling NJ. Post-operative neutrophil-lymphocyte ratio predicts complications following colorectal surgery. Int J Surg. 2007 Feb;5(1):27-30. doi: 10.1016/j.ijsu.2006.05.013. Epub 2006 Jun 27. PMID 17386911
- See also: CovidSurg Cohort Study. Globalsurg. — https://globalsurg.org/covidsurgcohortstudy/
- Available data/document: Individual Participant Data Set: 285260 — https://www.myresearchproject.org.uk/ — Data collection template available on IRAS (Integrated Research Application System) registration
- Available data/document: Statistical Analysis Plan: 285260 — https://www.myresearchproject.org.uk/ — Statistical analysis plan as part of protocol available on IRAS (Integrated Research Application System) registration
- Available data/document: Study Protocol: 285260 — https://www.myresearchproject.org.uk/ — Protocol available on IRAS (Integrated Research Application System) registration

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT04419571/Prot_SAP_000.pdf